CLINICAL TRIAL: NCT01296516
Title: Early Postpartum Treatment of Gestational Diabetes With Weight Loss and Exercise
Brief Title: Postpartum Weight Loss and Exercise (PRIDE)
Acronym: PRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: THE C.B. AND IRENE PENNINGTON FOUNDATION (Unknown)
Responsible Party: Principal Investigator, Leanne Redman, Principle Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: PBRC 10041
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Gestational Diabetes; Glucose Intolerance
Keywords: Women; Postpartum; GDM
MeSH Terms: conditions — Diabetes, Gestational; Glucose Intolerance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (Placebo Comparator): A group matched for age and BMI will be selected to serve as control subjects in this study.
  Interventions: Behavioral: Non-intervention group
- Face-to-face group (Active Comparator): Participants randomized to the face-to-face intervention will attend motivational meetings held once per week in Phase I and biweekly in Phase II. Behavioral sessions will be led by a trained interventionist and will take place at Pennington Biomedical Research Center.
  Interventions: Behavioral: Face to face
- Telehealth Group (Active Comparator): Participants randomized to the Telehealth intervention will receive behavioral counseling through Trestletree, phone system.
  Interventions: Behavioral: Telehelath Group

INTERVENTIONS:
Behavioral: Non-intervention group — A pedometer and written material on a healthy lifestyle.
  Other Names: Placebo
  Arms: Control Group
Behavioral: Face to face — Motivational meetings held once per week; Behavioral sessions weill be led by a trained interventionist.
  Arms: Face-to-face group
Behavioral: Telehelath Group — Participants will speak to Trestletree personnel once a week via phone.
  Other Names: Trestletree
  Arms: Telehealth Group

SUMMARY:
The overall objective of this pilot project is to test in 50 women with a history of gestational diabetes mellitus (GDM), the effectiveness and feasibility of an 8 month intensive lifestyle intervention to reduce the rate of metabolic abnormalities within 1 year after delivery.

DETAILED DESCRIPTION:
The objective is in comparison to a group of women not enrolled in the lifestyle intervention, 8 months of intensive lifestyle intervention aimed at promoting 7% weight loss through increased physical activity and dietary modification in women with a history of GDM will:

1. decrease body weight and
2. reduce the rate of metabolic abnormalities, 12 months after delivery

ELIGIBILITY:
Inclusion Criteria:

* Women are required to be enrolled (provided written consent for participation) in the COPSS-GDM study and therefore have met the following inclusion criteria:

  * Postpartum Women ≥18 years to 45 years (inclusive) of age who experienced GDM during index pregnancy
  * English-speaking

Exclusion Criteria:

* Exclusion Criteria:

  * Women enrolled in COPSS-GDM will be excluded if they met the following criteria:

Medical Exclusion Criteria

* History or clinical manifestation of any other significant metabolic, hematologic, pulmonary, cardiovascular, gastrointestinal, neurologic, immune, hepatic, renal, urologic disorders, or cancer
* Regular use of medications for weight control or psychosis
* Current use of medication to treat diabetes Psychiatric and Behavioral Exclusion Criteria
* History or clinical manifestation of any eating disorder
* Smoking
* History of drug or alcohol abuse (up to 14 drinks a week are allowed) within the past two years Other Exclusion Criteria
* Pregnancy or pregnancy planned during the coming year
* Unwilling or unable to adhere to the clinical evaluation schedule over the twelve -month study period

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2011-02; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Incidence of glucose intolerance | 8 Months
  To examine the incidence of glucose abnormalities (impaired fasting glucose, impaired glucose tolerance, type 2 diabetes) and health outcomes (changes in body fat, waist circumference and blood lipids)in women with a history of gestational diabetes, 12 months postpartum.

SECONDARY OUTCOMES:
Weight loss | 8 months
  Weight loss through increased physical activity and dietary modification will achieve similar results when delivered via face-to-face contact (DPP) or via telehealth

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M. Redman, PhD, Principal Investigator — Pennington Biomedical Research Center; Karen Elkind-Hirsh, PhD, Study Director — Womans' Research Hospital; Catherine Chamagne, PhD, Study Chair — Pennington Biomedical Research Center; Timothy S. Church, MD, MPH, PhD, Study Chair — Pennington Biomedical Research Center; Eric Ravussin, PhD, Study Chair — Pennington Biomedical Reserach Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States